CLINICAL TRIAL: NCT01961934
Title: Carbon-11-Sodium Acetate Positron Emission Tomography/Computed Tomography (PET/CT) Imaging Evaluation in Brain Glioma, Post Therapy Necrosis and Pseudo-progression
Brief Title: C11-Sodium Acetate PET/CT Imaging Evaluation in Brain Glioma, Post Therapy Necrosis and Pseudo-progression
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Awaiting funding
Sponsor: Phoenix Molecular Imaging (Other)
Responsible Party: Principal Investigator, Fabio Almeida MD, Medical Director/PI, Phoenix Molecular Imaging
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AMIC-AC-003
Record Dates: First submitted 2013-10-09; First posted 2013-10-14 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Gliomas
Keywords: glioblastoma; high grade brain tumors; recurrent; pseudo-progression; radionecrosis; carbon acetate; C11 aceate; PET; positron emission tomography
MeSH Terms: conditions — Glioma; Glioblastoma; Recurrence | interventions — Carbon-11; carbon-11 acetate; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sodium Acetate C11 PET/CT Imaging (Experimental)
  Interventions: Drug: Sodium Acetate C11 PET/CT Imaging

INTERVENTIONS:
Drug: Sodium Acetate C11 PET/CT Imaging
  Other Names: Carbon 11 Acetate; C11 Acetate; AC-PET; PET Imaging with Acetate C11

SUMMARY:
This study will investigate how well Carbon Acetate PET/CT imaging helps to correctly identify recurrent tumor versus post treatment effects (radionecrosis) in patients with previously treated high grade brain gliomas.

DETAILED DESCRIPTION:
The study is designed to investigate the effectiveness of Carbon Acetate PET/CT (AC PET)in terms of its ability to distinguish between radionecrosis/pseudo-progression and viable tumor in patients previously treated with surgery and radiation for high grade glioma brain tumors.

Eligible patients with biopsy proven high grade gliomas (WHO grades 3 and 4) status-post prior cranial irradiation for this tumor; age 18 to 70; ECOG/Zubrod of 0-2, no other contraindications to trial entry, and a post-irradiation cranial MRI or CT demonstrating an enhancing lesion of uncertain etiology (not biopsied) will be treated with at least two weeks of steroidal therapy.

Responders to steroidal therapy will be classified as either pseudo-progression (if asymptomatic) or radionecrosis (if symptomatic). Non-responders (those who do not respond clinically, radiographically, or both) will be referred for an FDG PET/CT and initial AC PET/CT within 3 weeks, and subsequently referred for stereotactic biopsy of their lesion followed by focal laser treatment (in the same operative setting) within 3 weeks of AC PET/CT.

Specific Goals/Questions:

1. What is the yield (sensitivity, accuracy, positive and negative predictive value) of state-of-the-art PET/CT with C-11 Acetate in detecting recurrent disease versus post treatment effects and pseudo-progression in this patient population?
2. How does the performance of PET with C-11 Acetate compare with that of PET using F-18 fluorodeoxyglucose (FDG-PET) and with that of MRI?
3. Evaluate the optimal timing for post injection imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18-70
* Pathologically confirmed World Health Organization (WHO) grade 3 or 4 glioma
* ECOG/Zubrod 0-2
* Prior external beam radiotherapy to 59.4-60 Gray by 1.8-2 Gy fractions
* Post-radiotherapy contrast-enhanced cranial MRI obtained at least 6 weeks after the completion of external beam radiotherapy shows enhancing anomaly (recurrent/progressive tumor versus pseudo-progression versus radionecrosis)
* Patient completed at least a two week course of palliative steroid therapy for this enhancing anomaly
* No prior designated therapy other than steroids for presumed radionecrosis or recurrent tumor
* Patient with no clinical and/or radiological response to steroid therapy
* Patient eligible for stereotactic brain biopsy
* Patient eligible for focal laser therapy

Exclusion Criteria:

* Patients under the age of 18 years
* Claustrophobic patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Biopsy Correlation | 3 weeks from AC PET Imaging
  AC PET imaging results will be correlated with tissue biopsy results

SECONDARY OUTCOMES:
SUV (Standardized Uptake Value) | Day 1 - Assess at time of PET imaging
  Imaging studies will be evaluated both qualitatively and quantitatively using SUV (standardized uptake values): a measure of metabolism based on injected dose, patient weight and region of interest. Comparison of the lesional activity to normal contralateral tracer activity will also be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Almeida, MD, Principal Investigator — Medical Director, Phoenix Molecular Imaging
Locations (1):
- Phoenix Molecular Imaging, Phoenix, Arizona, United States